CLINICAL TRIAL: NCT00000633
Title: A Phase I Multicenter Clinical Trial to Evaluate the Safety and Immunogenicity of Immuno-AG Recombinant HIV gp160 in Asymptomatic HIV Seropositive Individuals
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Immuno-US (Industry)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: ACTG 205; 11182 (Registry Identifier: DAIDS ES Registry Number); AVEG 101
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-02 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Vaccines, Synthetic; Vaccinia Virus; Viral Vaccines; HIV-1; HIV Envelope Protein gp160; Acquired Immunodeficiency Syndrome; AIDS-Related Complex; AIDS Vaccines; HIV Therapeutic Vaccine
MeSH Terms: conditions — HIV Infections; Vaccinia; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — Hepatitis B Vaccines

INTERVENTIONS:
Biological: gp160 Vaccine (Immuno-AG)
Biological: Hepatitis B Vaccine (Recombinant)

SUMMARY:
To determine the safety and immunogenicity of vaccinia-derived HIV-1 recombinant envelope glycoprotein (gp160) in asymptomatic HIV-infected adult volunteers. To compare safety and immunogenicity of two different schedules of gp160 administration. To examine the effects of gp160 and hepatitis B vaccine (Engerix-B) on various markers of viral load and on selected immune parameters.

Potentiation of a patient's immune response to HIV might possibly prolong the period of clinical latency and protect the patient indefinitely. Preliminary results from a study of Immuno-AG recombinant gp160 vaccine in healthy volunteers not infected with HIV suggest that the vaccine is safe and produces antibodies against the virus. Because another previous study failed to demonstrate a specific anti-HIV response in patients injected with a recombinant vaccinia virus containing HIV-1 genes, this study is also testing the immunotherapeutic role of other immunizations (such as hepatitis B vaccination) that would be expected to induce a nonspecific immune response in HIV-infected persons.

DETAILED DESCRIPTION:
Potentiation of a patient's immune response to HIV might possibly prolong the period of clinical latency and protect the patient indefinitely. Preliminary results from a study of Immuno-AG recombinant gp160 vaccine in healthy volunteers not infected with HIV suggest that the vaccine is safe and produces antibodies against the virus. Because another previous study failed to demonstrate a specific anti-HIV response in patients injected with a recombinant vaccinia virus containing HIV-1 genes, this study is also testing the immunotherapeutic role of other immunizations (such as hepatitis B vaccination) that would be expected to induce a nonspecific immune response in HIV-infected persons.

Fifty-five healthy HIV-positive volunteers are randomly assigned to one of the following treatment arms: six injections (arm I) or four injections (arm II) of HIV-1 gp160 vaccine, four injections of hepatitis B vaccine as a non-HIV viral vaccine control (arm III), or six placebo injections consisting of the adjuvant vehicle used for the gp160 vaccine (arm IV). Immunizations or placebo are given at 4-week intervals for 5 months. To maintain blinding, adjuvant vehicle placebo is administered on days 84 and 112 to those volunteers receiving four instead of six vaccine injections (arms II and III). Volunteers are followed at 4-month intervals for 2 years.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication: Recommended:

* Prophylaxis with isoniazid in patients not previously treated.

Patients must have:

* HIV seropositivity by Western blot.
* Normal history and physical exam (generalized lymphadenopathy is acceptable).
* Mean CD4 cell count = or > 600 cells/mm3 for all visits (minimum 2 counts) within 60 days prior to study entry, with no single count < 450 cells/mm3.
* Negative PPD test or normal chest x-ray with positive PPD (induration = or > 5 mm).

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Hepatitis B surface antigen positive.
* Evidence of an AIDS- or ARC-defining opportunistic infection.
* Evidence of disseminated tuberculosis, severe or persistent candidiasis, oral hairy leukoplakia, prolonged or very severe diarrhea, herpes zoster, or herpes simplex persisting more than one month.
* Active syphilis.

Patients with the following prior conditions are excluded:

* Evidence of psychiatric disorder within the past year that would impair adherence to the protocol.
* History of an AIDS- or ARC-defining opportunistic infection.
* History of disseminated tuberculosis, severe or persistent candidiasis, oral hairy leukoplakia, prolonged or very severe diarrhea, herpes zoster, or herpes simplex persisting more than one month.

Prior Medication:

Excluded:

* Immunomodulating agents (e.g., isoprinosine, imuthiol, lithium) within 90 days of screening.
* Immunosuppressive medications within the previous 3 months.
* Zidovudine (AZT) or any antiviral agent (including interferon) within the previous 6 months.
* Vaccination against other pathogens within 4 weeks of initial screening laboratory work.

Use of illicit drugs or significant amounts of alcohol that could significantly interfere with study compliance.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 55
Dates: Study Completion 1998-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Schwartz D, Study Chair
Locations (2):
- United States (2):
  - Johns Hopkins Adult AIDS CRS, Baltimore, Maryland
  - Washington U CRS, St Louis, Missouri

REFERENCES:
- [Background] Keefer MC, Graham BS, Belshe RB, Schwartz D, Corey L, Bolognesi DP, Stablein DM, Montefiori DC, McElrath MJ, Clements ML, et al. Studies of high doses of a human immunodeficiency virus type 1 recombinant glycoprotein 160 candidate vaccine in HIV type 1-seronegative humans. The AIDS Vaccine Clinical Trials Network. AIDS Res Hum Retroviruses. 1994 Dec;10(12):1713-23. doi: 10.1089/aid.1994.10.1713. PMID 7888231
- [Background] Belshe RB, Clements ML, Dolin R, Graham BS, McElrath J, Gorse GJ, Schwartz D, Keefer MC, Wright P, Corey L, et al. Safety and immunogenicity of a fully glycosylated recombinant gp160 human immunodeficiency virus type 1 vaccine in subjects at low risk of infection. National Institute of Allergy and Infectious Diseases AIDS Vaccine Evaluation Group Network. J Infect Dis. 1993 Dec;168(6):1387-95. doi: 10.1093/infdis/168.6.1387. PMID 8245523